CLINICAL TRIAL: NCT04166097
Title: Primary Prevention of Cardiovascular Disease Among Female Hospital Employees: The Heart Smart for Women Intervention
Acronym: Heart Smart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-0971
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Smart Interventional Program (Experimental): Subjects participate in this 6-week intervention which include a weekly didactic session, with each week devoted to a different theme (food, exercise, etc). The intervention will follow the program outlined in the book "Heart Smart for Women: Six S. T. E. P. S. in Six Weeks to Heart-Healthy Living."
  Interventions: Other: Heart Smart Interventional Program

INTERVENTIONS:
Other: Heart Smart Interventional Program — 6-week program consisting of weekly didactic sessions that follow the steps outlined in the book.

SUMMARY:
This study aims to show that a 6-week program designed specifically for women can lead to sustainable behavior change and improvement in heart disease risk factors over one year among a cohort of 46 female employees recruited from within the Heart Hospital at North Shore University Hospital (NSUH). The program is adapted from book "Heart Smart for Women: Six S. T. E. P. S in Six Weeks to Heart-Healthy Living," written by Northwell cardiologists Dr. Jennifer H. Mieres and Dr. Stacey E. Rosen.

The 6-week intervention will include a weekly didactic session, with each week devoted to a different theme (food, exercise, etc). The intervention will follow the program outlined in the book. We will also be using Yammer, an online discussion group part of the Office 365 suite, to distribute materials and encourage conversations surrounding the theme of the week.

DETAILED DESCRIPTION:
Heart Disease is the leading cause of death in women in the United State. Nine out of ten women have one or more risk factors for heart disease and one in three women will die of heart disease. However, most women are unaware of these statistics. As a result, women are less likely than men to recognize the symptoms of a heart attack and are more likely than men to delay in seeking help. The best ways to educate women about heart disease and change their behavior to prevent heart disease are unknown.

More than 80% of heart disease is preventable but requires both knowledge of risk factors and adherence to lifestyle changes. This program is designed to address these challenges in women, where this is a particular unmet need.

Some prior community and workplace-based studies have demonstrated short term improvements in modifiable risk factors for cardiovascular disease. A community based primary prevention program among disadvantaged women decreased the rate of metabolic syndrome, anxiety, depression and stress.

The economic burden of heart disease on employers is significant although workplace employee wellness programs have not been shown to decrease employer costs. The impact of employee wellness programs on clinical outcome measures have been inconsistent.

This program is designed to educate female employees about their heart disease risk factors and provide tactical support to improve their heart health. Once validated, the program can be rolled out to other employees and to the community.

ELIGIBILITY:
Inclusion Criteria:

* one or more of the following modifiable risk factors for cardiovascular disease [as defined by the American Heart Association]:

  1. cigarette smoking
  2. high blood pressure
  3. high cholesterol
  4. abnormal blood sugar
  5. sedentary lifestyle
  6. overweight/obese
* must be an employee of the Heart Hospital at North Shore University Hospital

Exclusion Criteria:

* prior history of heart attack or stroke
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Decreased Blood Pressure | 1 year
  Blood Pressure at a single follow-up measured as 2 readings separated by 5 minutes. This will be observed at baseline, end of 6-week program, 3 months post-completion, 6 months post-completion, and 1 year post-completion.
  Significant change in this outcome will be defined as a difference in means of 7 mmHg between baseline average and follow-up average.
Decreased Total Cholesterol | 1 year
  Total Cholesterol measured by lipid profile of blood drawn. This will be observed at baseline, end of 6-week program, 3 months post-completion, 6 months post-completion, and 1 year post-completion.
Decreased Low Density Lipoprotein Cholesterol (LDL-C) | 1 year
  Low Density Lipoprotein Cholesterol (LDL-C) measured by lipid profile of blood drawn. This will be observed at baseline, end of 6-week program, 3 months post-completion, 6 months post-completion, and 1 year post-completion.
Decreased Body Mass Index (BMI) | 1 year
  Weight in kilograms and height in meters will be combined to report BMI in kg/m^2. This will be observed at baseline, end of 6-week program, 3 months post-completion, 6 months post-completion, and 1 year post-completion.
Decreased Waist Circumference | 1 year
  This will be observed at baseline, end of 6-week program, 3 months post-completion, 6 months post-completion, and 1 year post-completion.

SECONDARY OUTCOMES:
Decreased HbA1c | 1 year
Decreased Psychosocial Stress | 1 year
  Psychosocial Stress scored via the Perceived Stress Scale (PSS). The minimum value is 0 and the maximum value is 40, with higher scores meaning worse outcome.
Decreased Depression Score | 1 year
  Depression scored via Patient Health Questionnaire-4 (PHQ-4). The minimum value is 0 and the maximum value, with higher scores meaning worse outcome. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
Decreased Sleep Disturbance | 1 year
  Sleep Disturbance scored via Pittsburgh Sleep Quality Index (PSQI). The minimum value is 0 and the maximum value is 21, with higher scores meaning worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey E Rosen, MD, Principal Investigator — Northwell Health; Katz Women's Hospital at Long Island Jewish Medical Center
Locations (1):
- Sandra Atlas Bass Heart Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI has identified an independent data and safety monitor, Dr. Penny Stern, who has expertise in cardiovascular prevention and who does not have any scientific, financial, or other conflict of interest related to the study and who is not responsible for patient care at any of the participating sites.
  Study protocol will be reviewed and record keeping done every 3 months to ensure that all employee/participant information is kept confidential.
  Password-protected database will be used to enter all data - it will contain only de-identified information. Moreover, the online discussion group, Yammer, activity will be reviewed to ensure participant confidentiality is maintained and that unauthorized disclosure of information outside the private group is prevented.
Supporting Information: Study Protocol, CSR
Time Frame: Data available: January 2020 Duration available: 1 year, 1 month

REFERENCES:
- [Background] Gilstrap LG, Malhotra R, Peltier-Saxe D, Slicas D, Pineda E, Culhane-Hermann C, Cook N, Fernandez-Golarz C, Wood M. Community-based primary prevention programs decrease the rate of metabolic syndrome among socioeconomically disadvantaged women. J Womens Health (Larchmt). 2013 Apr;22(4):322-9. doi: 10.1089/jwh.2012.3854. Epub 2013 Mar 29. PMID 23540328
- [Background] Thorndike AN. Workplace Interventions to Reduce Obesity and Cardiometabolic Risk. Curr Cardiovasc Risk Rep. 2011 Feb;5(1):79-85. doi: 10.1007/s12170-010-0138-0. PMID 22708000
- [Background] Kim DA, Hwong AR, Stafford D, Hughes DA, O'Malley AJ, Fowler JH, Christakis NA. Social network targeting to maximise population behaviour change: a cluster randomised controlled trial. Lancet. 2015 Jul 11;386(9989):145-53. doi: 10.1016/S0140-6736(15)60095-2. Epub 2015 May 4. PMID 25952354
- [Background] Riegel B, Moser DK, Buck HG, Dickson VV, Dunbar SB, Lee CS, Lennie TA, Lindenfeld J, Mitchell JE, Treat-Jacobson DJ, Webber DE; American Heart Association Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; and Council on Quality of Care and Outcomes Research. Self-Care for the Prevention and Management of Cardiovascular Disease and Stroke: A Scientific Statement for Healthcare Professionals From the American Heart Association. J Am Heart Assoc. 2017 Aug 31;6(9):e006997. doi: 10.1161/JAHA.117.006997. PMID 28860232
- [Background] Thorndike AN, Healey E, Sonnenberg L, Regan S. Participation and cardiovascular risk reduction in a voluntary worksite nutrition and physical activity program. Prev Med. 2011 Feb;52(2):164-6. doi: 10.1016/j.ypmed.2010.11.023. Epub 2010 Dec 3. PMID 21130804
- [Background] Richardson G, van Woerden HC, Morgan L, Edwards R, Harries M, Hancock E, Sroczynsk S, Bowley M. Healthy hearts--a community-based primary prevention programme to reduce coronary heart disease. BMC Cardiovasc Disord. 2008 Jul 26;8:18. doi: 10.1186/1471-2261-8-18. PMID 18655720
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Sep 10;74(10):1376-1414. doi: 10.1016/j.jacc.2019.03.009. Epub 2019 Mar 17. PMID 30894319
- [Background] Makaryus AN, Rosen SE, Kang L, Shaw LJ, Nash B, Gajer R, Coppolino W, Mieres JH. Racial and Ethnic Differences in Awareness and Prevalence of Unidentified Cardiovascular Risk Factors Among Health System Employees. Am J Health Promot. 2023 Nov;37(8):1091-1099. doi: 10.1177/08901171231192484. Epub 2023 Jul 26. PMID 37492930